CLINICAL TRIAL: NCT07300293
Title: Prognosis of Lactic Acidosis Upon Admission to Intensive Care According to the Existence of Prior Treatment With Metformin
Brief Title: Lactic Acidosis and Prior Metformin Treatment
Acronym: MALA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9381
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Metformin Treatment; Lactic acidosis; Metabolic acidosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Acidosis, Lactic; Acidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metformin is a drug frequently prescribed to patients with type 2 diabetes. Furthermore, diabetes can lead to micro- and macrovascular complications that may cause chronic organ failure. The presence of diabetes also increases the risk of infections. All of these factors contribute to the frequent admission of patients to the ICU who have been receiving metformin treatment in the preceding days. Acute renal failure, which is also frequently observed upon admission to the ICU, increases the risk of metformin overdose. In cases of overdose, metformin acts on several metabolic pathways that can lead to or even accelerate metabolic acidosis, sometimes severe. However, the impact on prognosis is controversial.

The role of metformin in lactic acidosis in patients treated for acute illness may be underestimated in routine practice.

This study aims to investigate the impact of prior metformin treatment on ICU survival in patients admitted to the ICU with severe lactic acidosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years)
* Admitted to the intensive care unit of Hautepierre Hospital - Strasbourg University Hospital between January 1, 2014, and December 31, 2023
* Having experienced lactic acidosis (pH <7.35 and lactate level ≥5 mmol/L) within the first 24 hours of hospitalization.

Exclusion Criteria:

* Patient without arterial blood gas measurements during the first 24 hours of admission
* whose background treatment is unknown and could not be determined
* for whom a limitation of active therapies was implemented before or during the first 24 hours of hospitalization

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years) having experienced lactic acidosis (pH <7.35 and lactate level ≥5 mmol/L) within the first 24 hours of hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Survival rates of patients with severe lactic acidosis admitted to the ICU after prior metformin treatment | Up to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Intensive - Réanimation - CHU de Strasbourg - France, Strasbourg, France